CLINICAL TRIAL: NCT07180472
Title: Prevention of Stroke Recurrence and Disease Progression in Cerebral Small Vessel Disease With Cilostazol: a Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Prevention of Stroke Recurrence and Disease Progression in Cerebral Small Vessel Disease With Cilostazol
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025CYFYIRB-BA-113
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Small Vessel Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Cilostazol; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol group (Experimental)
  Interventions: Drug: Cilostazol
- Orignal threapy group (Active Comparator): Asprin or clopidogrel
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cilostazol — Oral administration of cilostazol
  Arms: Cilostazol group
Drug: Aspirin — Oral administration of Asprin
  Arms: Orignal threapy group
Drug: Clopidogrel — Oral administration of Clopidogrel
  Arms: Orignal threapy group

SUMMARY:
This study is designed to evaluate whether cilostazol, an antiplatelet medication, is more effective and safer than aspirin or clopidogrel in preventing recurrent strokes and slowing disease progression in patients with cerebral small vessel disease (CSVD).

Cerebral small vessel disease is a common cause of lacunar stroke, cognitive decline, and long-term disability. Currently, aspirin and clopidogrel are widely used to prevent recurrent ischemic events, but their effectiveness in CSVD remains uncertain. Cilostazol has shown potential benefits in improving cerebral blood flow, protecting blood vessel walls, and reducing the risk of bleeding compared with traditional antiplatelet drugs.

In this randomized controlled trial, participants diagnosed with CSVD and recent lacunar stroke will be randomly assigned to receive cilostazol, aspirin, or clopidogrel. The main outcomes to be evaluated include the rate of recurrent ischemic stroke, progression of cognitive and functional impairment, MRI markers of CSVD (such as white matter hyperintensity, lacunes, microbleeds, and small infarcts), and safety outcomes including bleeding events.

The investigators hypothesize that cilostazol will reduce the risk of recurrent stroke and slow disease progression more effectively than aspirin or clopidogrel, with a comparable or lower risk of bleeding.

By comparing these three antiplatelet drugs in a rigorous, multicenter randomized controlled trial, this study will provide important clinical evidence to guide personalized treatment strategies for patients with CSVD. The results are expected to improve long-term outcomes, reduce disability, and enhance the quality of life for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Diagnosis of small artery occlusion ischemic stroke based on the TOAST classification, with symptom onset within the past 6 months.
3. MRI findings indicating white matter hyperintensities, with Fazekas grade ≥2.
4. mRS (modified Rankin Scale) score ≤2.
5. CDR (Clinical Dementia Rating) score <1.

Exclusion Criteria:

1. Presence of other central nervous system (CNS) disorders, including CNS infections, immune-mediated or degenerative diseases, epilepsy, intracranial tumors, etc.
2. History of drug or alcohol abuse, or severe psychiatric disorders.
3. Diagnosis of malignant tumors.
4. Severe hepatic dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3 times the upper limit of normal) or renal impairment (creatinine clearance <25 mL/min).
5. Concomitant congestive heart failure.
6. Systemic hemorrhagic disorders or bleeding tendency, including platelet count ≤100,000/mm³, coagulation abnormalities, gastrointestinal ulcers, or history of non-traumatic symptomatic intracranial hemorrhage.
7. Conditions requiring long-term anticoagulation therapy, such as atrial fibrillation or deep vein thrombosis.
8. Known allergy or contraindication to cilostazol, clopidogrel, or aspirin.
9. Requirement for dual antiplatelet therapy during the study period (e.g., due to vascular stent implantation or symptomatic intracranial arterial stenosis).
10. Inability to complete scale assessments or comply with long-term follow-up.
11. Pregnancy, lactation, or planning to become pregnant.
12. Participation in another interventional clinical trial.
13. Any other condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of composite events, including new-onset ischemic stroke, transient ischemic attack, cognitive impairment, functional disability, and death | Day 360

IPD SHARING:
Plan to Share IPD: No